CLINICAL TRIAL: NCT02785601
Title: Pharmacokinetics Study of Trazodone Hydrochloride Prolonged -Released Tablets in Chinese Healthy Volunteers
Brief Title: PK Study of Diet Effect of Trazodone Hydrochloride Prolonged-Released Tablets in Healthy Chinese
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: Zhaoke-201603-Tra-Trial I
Record Dates: First submitted 2016-05-24; First posted 2016-05-30 (Estimated); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- I-1 (Experimental): This is a four different crossover treatments with 2 men and 2 women, give the following treatment sequence, with wash out period 7 days (A) postprandial single oral dose of trazodone hydrochloride prolonged-release tablets 75 mg; (D) postprandial single oral trazodone hydrochloride tablets 150mg (50mg for 3 times) (B) postprandial single oral dose of trazodone hydrochloride prolonged-release tablets 150 mg; (C) fasting single oral dose of trazodone hydrochloride prolonged-release tablets 150 mg;
  Interventions: Drug: Trazodone Hydrochloride prolonged-release tablets
- I-2 (Experimental): This is a four different crossover treatments with 2 men and 2 women, give the following treatment sequence, with wash out period 7 days (B) postprandial single oral dose of trazodone hydrochloride prolonged-release tablets 150 mg; (A) postprandial single oral dose of trazodone hydrochloride prolonged-release tablets 75 mg; (C) fasting single oral dose of trazodone hydrochloride prolonged-release tablets 150 mg; (D) postprandial single oral trazodone hydrochloride tablets 150mg (50mg for 3 times)
  Interventions: Drug: Trazodone Hydrochloride prolonged-release tablets
- I-3 (Experimental): This is a four different crossover treatments with 2 men and 2 women, give the following treatment sequence, with wash out period 7 days (C) fasting single oral dose of trazodone hydrochloride prolonged-release tablets 150 mg; (B) postprandial single oral dose of trazodone hydrochloride prolonged-release tablets 150 mg; (D) postprandial single oral trazodone hydrochloride tablets 150mg (50mg for 3 times) (A) postprandial single oral dose of trazodone hydrochloride prolonged-release tablets 75 mg;
  Interventions: Drug: Trazodone Hydrochloride prolonged-release tablets
- I-4 (Experimental): This is a four different crossover treatments with 2 men and 2 women, give the following treatment sequence, with wash out period 7 days (D) postprandial single oral trazodone hydrochloride tablets 150mg (50mg for 3 times) (C) fasting single oral dose of trazodone hydrochloride prolonged-release tablets 150 mg; (A) postprandial single oral dose of trazodone hydrochloride prolonged-release tablets 75 mg; (B) postprandial single oral dose of trazodone hydrochloride prolonged-release tablets 150 mg;
  Interventions: Drug: Trazodone Hydrochloride prolonged-release tablets

INTERVENTIONS:
Drug: Trazodone Hydrochloride prolonged-release tablets — strength 75mg, 150 mg. Oral administration with 200ml water

SUMMARY:
The main objective is to compare the pharmacokinetics in single dose, and effect of food on the trazodone hydrochloride pharmacokinetics prolonged-release tablets.

DETAILED DESCRIPTION:
Trial I single dose (75mg and 150mg), fasting or postprandial comparative pharmacokinetics of trazodone hydrochloride prolonged-release tablets and ordinary formulation; 16 patients (males and females, half and half).

Trial is a 4-period, 4 cross (4x4) Williams crossover design, screened 16 subjects (half males and half females) were randomly divided into four groups (I-1, I-2, I-3, I-4), each 2 men and 2 women, give the following four different crossover treatments:

(A) postprandial single oral dose of trazodone hydrochloride prolonged-release tablets 75 mg; (B) postprandial single oral dose of trazodone hydrochloride prolonged-release tablets 150 mg; (C) fasting single oral dose of trazodone hydrochloride prolonged-release tablets 150 mg; (D) postprandial single oral trazodone hydrochloride tablets 150mg (50mg for 3 times) Time for drug administration is around 8:00am. Wash-out period is 7 days. Blood sampling will be performed before (0h) and after administration each dose group 0.5, 1.0, 2.0, 3.0, 4.0, 5.0, 6.0, 8.0, 10.0, 12.0, 16.0, 24.0, 36.0, 48.0, 72.0h.

Trial I. 4X4 Williams design Group Period 1 Period 2 Period 3 Period 4 I-1 A D B C I-2 B A C D I-3 C B D A I-4 D C A B

ELIGIBILITY:
Inclusion Criteria:

* Weight: all the subjects should be ≥50 kg, BMI within 19~24 kg/m2；
* Blood pressure: SBP 90-140mmHg，DBP 50-90 mmHg；
* All the subjects should understand this trial well and sign the inform consent form before participating this study;
* Subjects should be able to communicate with investigators well and complete this study in accordance with protocol.

Exclusion Criteria:

* The baseline value of safety evaluation index is considered to be abnormal with clinical significance by investigators before participating the trial.
* A positive hepatitis B surface antigen result；
* A positive hepatitis C surface antigen result；
* A positive test for HIV antibody and syphilis testing；

Any of the abnormalities of ECGs examination occurs in screening period or the first day of administration:

* With the history of using any drug which will inhibit or induce liver to metabolize drug within 1 month before the study initiation;
* With the history of administrating any drugs (prescription medicine, over-the-counter drug and Chinese herbal medicine) within 2 week before the study initiation;
* Past history of heart disease, cardiac failure, myocardial infarction, angina, unknown cause of arrhythmia, point swinging pattern of ventricular tachycardia, ventricular tachycardia, long QT syndrome or long QT syndrome and family history (with genetic proof or there were any close relatives died because of heart disease);
* History of thyroid disease or past history of thyroid surgery;
* History of immune system disease (such as thymus disease)；
* With surgery history within 6 months before this study initiation；
* History of severe digestive disease (such as gallbladder disease with significant clinical significance, jaundice or susceptive jaundice, hepatocellular adenoma, hepatic cavernous hemangioma and the other liver diseases)；
* With history of gastrointestinal, liver and renal disease (no matter it has been cured or not) which will affect drug absorption and metabolism within 6 months before this study initiating；
* History of any serve cardiocerebral vascular system, respiratory system, metabolic system and nervous system diseases;
* History of hematological system diseases, such as coagulation disorders；
* History of tumor；
* Subjects with hypokalemia and hypocalcemia (according to the lower limit value of the laboratory reference ranges；

Life style:

* History of alcohol addicted within 6 months before the study
* Smoking >1 cigarettes a day in the last 3 months prior to this study;
* History of drug abuse and taking drugs (such as marihuana, cocaine, opium, benzodizepines, amphetamines, barbiturates, tricyclic antidepressant).
* History of consumption of excessive tea, coffee and/or caffeinated beverage (more than 8 cups/day) within the period of 2 days before the administration and 8 days after administration.
* History of consumption of grapefruit juice within the period of 2 days before and 8 days after administration.

Others：

* Subjects who reject to take effective contraceptive measures within the time period after inclusion to 3 months after administration;
* Subjects with allergic constitution, including those who are allergic to the excipient (microcrystalline cellulose, lactose, aerosil, sodium carboxymethyl starch, magnesium stearate) of this product;
* History of participating any clinical trial within 3 months before this study, or participating the other clinical trial within the time period of inclusion to one month after the last time visit(after the last time administration);
* History of blood donation within 3 months prior to this study, or within the time period of inclusion to one month after the last time visit (after the last time administration);
* Subjects who have food allergy or have any special diet requirements, or who cannot follow the standard diet;
* Subjects who, in the opinion of the investigator, should not participate in the study.

The female subjects are not eligible for inclusion in this study if she meet any of the following criteria above and below:

* With the history of consumption of oral contraceptive within one month prior to this study；
* History of long-acting estrogen or progesterone injection or implant within 6 months prior to this study;
* The bearing-age female subjects who have not taken appropriate contraceptives within 2 weeks prior to this study;
* The bearing-age female subjects and their spouse are not willing to take the following contraceptives measure, condom, copper intrauterine device within 3 months after inclusion;
* Subjects who are in gestation period and lactation period;
* Subjects with positive hCG test;
* Single menstrual more than 80ml.

Ages: 19 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2017-05-01 (Actual); Primary Completion 2017-11-30 (Actual); Study Completion 2018-01-04 (Actual)

PRIMARY OUTCOMES:
Area Under Curve (AUC) | pre-dose, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 16 hours, 24 hours, 36 hours, 48 hours, 72 hours after administration
  To observe area under curve characteristics of trazodone hydrochloride prolonged-release tablets in single or multiple dose groups
Area Under Curve (AUC) | pre-dose, 30 minutes, 1 hour, 2 hours, 3 hours, 4 hours, 5 hours, 6 hours, 8 hours, 10 hours, 12 hours, 16 hours, 24 hours, 36 hours, 48 hours, 72 hours after administration
  To observe area under curve characteristics of trazodone hydrochloride prolonged-release tablets in fasting or high-fat diet groups

CONTACTS AND LOCATIONS:
Overall Officials: Andrea On Yan Luk, Principal Investigator — Prince of Wales Hospital
Locations (1):
- Prince of Wales Hospital, Hong Kong, Hong Kong